CLINICAL TRIAL: NCT07309744
Title: Clinical Study on Safety, Efficacy, and Pharmacokinetics of Universal CAR-T Cell Injection Targeting CD19/BCMA in Patients With Inflammatory Bowel Disease
Brief Title: Universal CAR-T Cell Injection Targeting CD19/BCMA in Patients With Inflammatory Bowel Disease
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BHCT-RD06-05-IBD
Record Dates: First submitted 2025-12-02; First posted 2025-12-30 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Moderate-to-severe Ulcerative Colitis; Crohn's Disease (CD)
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Intervention Model Description: This is an open-label, single-arm clinical study, in which all enrolled patients will receive the infusion of RD06-05 cell infusion.
  Two cohorts are established in the study to explore the optimal biological dose (OBD) for each indication:
  Cohort 1: Ulcerative Colitis Cohort Cohort 2: Crohn's Disease Cohort The study presets 3 dose groups, which are 3, 6, and 10×10⁶ CAR+T cells/kg respectively. The initial dose group is 3×10⁶ CAR+T cells/kg (Dose Group 1), and dose de-escalation or escalation may be conducted based on the assessment of the Safety Review Committee (SRC).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CART Treatment Group (Experimental): In this group, participants will receive the infusion of RD06-05 cell injection.
  Interventions: Drug: RD06-05 CART Cell Infusion

INTERVENTIONS:
Drug: RD06-05 CART Cell Infusion — Participent will receive the infusion of RD06-05 cell injection with dosage of 3, 6, or 10×10⁶ CAR+T cells/kg respectively

SUMMARY:
This is an open-label, Phase I, investigator-initiated trial (IIT) designed to evaluate the safety, tolerability, pharmacokinetics, pharmacodynamics, and efficacy of RD06-05 in patients with moderate-to-severe ulcerative colitis (UC) and Crohn's disease (CD). The enrolled population consists of patients with refractory moderate-to-severe inflammatory bowel disease who have received multiple lines of biologic therapy.

Two cohorts are established in the study to explore the optimal biological dose (OBD) for each indication:

Cohort 1: Ulcerative Colitis Cohort Cohort 2: Crohn's Disease Cohort The study presets 3 dose groups, which are 3, 6, and 10×10⁶ CAR+T cells/kg respectively. The initial dose group is 3×10⁶ CAR+T cells/kg (Dose Group 1), and dose de-escalation or escalation may be conducted based on the assessment of the Safety Review Committee (SRC).

It is expected that no more than 9 patients will be enrolled in each cohort.

ELIGIBILITY:
Inclusion Criteria:

* The subject voluntarily participates in this trial and signs the informed consent form.
* Aged ≥ 18 years and ≤ 70 years, regardless of gender.
* Organ function and laboratory tests:

  1. Liver function: Alanine Aminotransferase (ALT) and Aspartate Aminotransferase (AST) ≤ 2 × Upper Limit of Normal (ULN); Total Bilirubin (TBIL) ≤ 2 × ULN (except for Gilbert's syndrome).
  2. Renal function: Creatinine ≤ 1.5 × ULN or Creatinine Clearance ≥ 40 ml/min.
  3. Complete blood count: Neutrophil count ≥ 1 × 10⁹/L; Hemoglobin ≥ 60 g/L; Platelet count ≥ 20 × 10⁹/L; Lymphocyte count > 0.3 × 10⁹/L.
  4. Coagulation function: International Normalized Ratio (INR) ≤ 1.5 × ULN, or Prothrombin Time (PT) ≤ 1.5 × ULN.
  5. Oxygen saturation (SpO₂) ≥ 92% in room air at rest.
  6. Echocardiography shows Left Ventricular Ejection Fraction (LVEF) ≥ 50%.
* Female subjects of childbearing potential must have a negative result in serum or urine pregnancy test at screening.
* Female subjects of childbearing potential must agree to use highly effective contraceptive methods from at least 28 days before the start of lymphodepletion until 12 months after RD06-05 infusion. Male subjects of childbearing potential must agree to use effective barrier contraceptive methods from the start of lymphodepletion until 12 months after RD06-05 infusion, and must not donate semen or sperm during the entire trial period.

Inclusion Criteria for Patients with Ulcerative Colitis (UC)

* Diagnosis of ulcerative colitis confirmed by clinical and endoscopic evidence at least 3 months before screening, and verified by histopathological report. If no pathological report is available, additional biopsies may be performed during the screening period to obtain specimens, which will be sent to a local pathological laboratory for diagnostic confirmation.
* Moderate to severe active ulcerative colitis, defined as a Mayo score between 6 and 12 points with an endoscopic subscore ≥ 2 points (endoscopic examination performed within 14 days before screening).
* Confirmed that the extent of ulcerative colitis lesions involves above the rectosigmoid junction (approximately ≥ 15 cm from the anal verge).
* Patients with extensive colitis or pancolitis with a disease duration of more than 8 years, or left-sided colitis with a disease duration of more than 12 years, must have written evidence of having undergone a colonoscopy within 12 months before the first screening visit (may be performed during the screening period or within 14 days before screening).
* Subjects with a family history of colorectal cancer, personal history of high risk for colorectal cancer, age > 50 years, or other known risk factors must have completed colorectal cancer-related screening (including but not limited to colonoscopic biopsy, imaging, biomarkers, etc., which may be performed during the screening period).
* Previous proven inadequate response, loss of response, or intolerance to at least one of the following drugs:

Glucocorticoids:

After at least one cycle of induction therapy (equivalent to oral prednisone 30 mg daily for 2 weeks or intravenous administration for 1 week), signs and symptoms of persistent active disease still exist; OR Previous failure of at least two attempts to reduce glucocorticoid dosage to below oral prednisone 10 mg/day or equivalent dose; OR Previous history of glucocorticoid intolerance (including but not limited to: Cushing's syndrome, osteopenia or osteoporosis, hyperglycemia, insomnia, infection, etc.).

Immunomodulators:

After previous treatment with oral azathioprine (≥ 1.5 mg/kg) or 6-mercaptopurine (≥ 0.75 mg/kg) for at least 8 weeks, signs and symptoms of persistent active disease still exist; OR Previous history of intolerance to at least one immunomodulator (including but not limited to: nausea, vomiting, abdominal pain, pancreatitis, abnormal liver function tests, lymphopenia, TPMT gene mutation, infection, etc.).

* Patients with previous inadequate response, loss of efficacy, or intolerance to at least two drugs of different mechanism classes among biological therapy (such as anti-TNF antibodies, anti-IL antibodies, or anti-integrin antibodies) or Janus kinase (JAK) inhibitor therapy (such as upadacitinib) for ulcerative colitis. The aforementioned drugs must be domestically approved for the treatment of ulcerative colitis. Investigators must be able to provide relevant records of sufficient clinical treatment with the drug. Patients must meet any of the following criteria:

Inadequate efficacy: Despite induction therapy with the approved induction dose as specified in the drug instruction manual, the patient still shows signs and symptoms of persistent active disease; OR Loss of efficacy: On the basis of previous benefit, recurrence of signs and symptoms of active disease occurs during treatment with the approved maintenance dose as specified in the drug instruction manual (even if the drug is discontinued voluntarily after obtaining clinical benefit, it is not considered as biological therapy failure or intolerance to ulcerative colitis treatment); OR Intolerance: Previous history of intolerance to biological agents or JAK inhibitors approved for ulcerative colitis, including but not limited to infliximab, adalimumab, golimumab, ustekinumab, vedolizumab, upadacitinib, or others (including but not limited to infusion-related events, demyelination, congestive heart failure, or any drug-related adverse event leading to dose reduction or discontinuation).

* The following drugs are allowed to be used in the study under stable dosage:

Oral 5-aminosalicylic acid (5-ASA) treatment: The prescribed dosage has been used stably for at least 2 weeks before the screening colonoscopy; Oral glucocorticoid treatment (prednisone ≤ 20 mg/day or equivalent dose, or extended-release budesonide tablets 9 mg/day): The prescribed dosage has been used stably for at least 2 weeks before the screening colonoscopy.

* Having the condition to discontinue other therapeutic drugs for UC (except the above-mentioned allowed concomitant drugs) before pretreatment. For specific drugs, please refer to the "Section 7.14 Prohibited Concomitant Treatments" in the protocol and the corresponding drug washout period regulations.
* Willing and able to complete the scheduled study assessments, including but not limited to endoscopic examinations.

Inclusion Criteria for Patients with Crohn's Disease (CD)

* The subject must be diagnosed with Crohn's disease at least 3 months before enrollment, and the diagnosis must be confirmed by clinical, endoscopic, and histopathological criteria. If no pathological report is available, the investigator may obtain specimens through additional biopsies during the screening period and send them to a local pathological laboratory for diagnostic confirmation.
* The subject must be a patient with moderate to severe active Crohn's disease, defined as a Crohn's Disease Activity Index (CDAI) score ≥ 220 points during the screening period, and meet any of the following conditions:

Elevated C-reactive protein (CRP) level during the screening period (based on the upper limit of the reference range of the laboratory of each study center); OR Colonoscopy within 4 months before screening shows at least 3 non-anastomotic ulcers (each with a diameter > 0.5 cm) or at least 10 aphthous ulcers (involving a continuous intestinal segment ≥ 10 cm), consistent with the characteristics of Crohn's disease; OR Computed Tomography Enterography (CTE), Magnetic Resonance Enterography (MRE), Contrast-Enhanced Small Bowel Radiography, or Capsule Endoscopy within 4 months before screening shows Crohn's disease-related ulcers (patients with only aphthous ulcers, fixed strictures, or small bowel strictures with pre-stenotic dilatation should not be enrolled).

* Subjects with a family history of colorectal cancer, personal history of high risk for colorectal cancer, age > 50 years, or other known high-risk factors must complete the latest colorectal cancer monitoring (including but not limited to colonoscopy and endoscopic biopsy, imaging, tumor biomarkers, etc.).
* The subject has inadequate efficacy, loss of efficacy, or poor tolerance to at least one of the following drugs:

Glucocorticoids:

Glucocorticoid-refractory disease: Refers to subjects who still have signs and/or symptoms of active Crohn's disease after receiving oral prednisone (or equivalent drug) at a daily dose of ≥ 30 mg or budesonide at a daily dose of ≥ 9 mg for at least 4 weeks; OR Glucocorticoid-dependent disease: Refers to (1) inability to reduce the dose to prednisone equivalent dose < 10 mg/day or budesonide < 3 mg/day within 3 months after starting glucocorticoid use; or (2) recurrence within 3 months after completing a course of glucocorticoid treatment; OR Glucocorticoid intolerance: Refers to adverse reactions that lead to drug discontinuation when the subject uses glucocorticoids, including but not limited to Cushing's syndrome, osteopenia/osteoporosis, hyperglycemia, neuropsychiatric adverse reactions, etc.

Immunomodulators:

Persistent signs and/or symptoms of active disease still exist after using any of the following drugs for at least 3 months:

1. Oral azathioprine (AZA) at a daily dose of ≥ 1.5 mg/kg, or 6-mercaptopurine (6-MP) at a daily dose of ≥ 0.75 mg/kg, or methotrexate (MTX) at 25 mg per week (intramuscular injection or subcutaneous injection); OR
2. Oral AZA or 6-MP within the therapeutic range determined by thiopurine metabolite detection; OR
3. Combined use of thiopurine and allopurinol, and within the therapeutic range determined by thiopurine metabolite detection; OR Intolerance to at least one immunomodulator: Adverse reactions leading to drug discontinuation when using any immunomodulator, including but not limited to nausea/vomiting, abdominal pain, pancreatitis, abnormal liver function, lymphopenia.

   * Subject with biological therapy failure: Refers to subjects with inadequate efficacy, loss of efficacy, or poor tolerance to at least two biological agents of different mechanisms that have been approved for the treatment of Crohn's disease (such as anti-TNF antibodies, anti-IL antibodies, or anti-integrin antibodies). Investigators must be able to provide sufficient medication history records during the induction period and/or maintenance period. The subject must meet one of the following criteria:

Inadequate efficacy: Refers to persistent signs and/or symptoms of active disease after induction therapy with the induction dose specified in the product instruction manual; OR Loss of efficacy: Refers to the recurrence of signs and/or symptoms of active disease after obtaining clinical improvement during treatment with the approved maintenance dose; OR Poor tolerance: Refers to adverse reactions that lead to dose reduction or discontinuation when the subject uses domestically or approved biological agents (including but not limited to infusion-related events, demyelination, congestive heart failure, etc.).

* Subjects are allowed to use the following drugs concomitantly at a stable dose during the study:

Oral 5-aminosalicylic acid (5-ASA) treatment: The dose has been stable for at least 2 weeks before the screening colonoscopy; Oral glucocorticoid treatment (prednisone ≤ 20 mg/day or equivalent dose, or budesonide ≤ 9 mg/day): The dose has been stable for at least 2 weeks before the screening colonoscopy; Antibiotics specifically used for the treatment of Crohn's disease: If used continuously, the dose has been stable for at least 2 weeks before the screening colonoscopy; Probiotics: Such as Saccharomyces boulardii, etc., with a stable dose for at least 2 weeks before the screening colonoscopy; Antidiarrheals: Such as loperamide, compound diphenoxylate with atropine, etc., used to control chronic diarrhea.

* Having the condition to discontinue other therapeutic drugs for CD (except the above-mentioned allowed concomitant drugs) before pretreatment. For specific drugs, please refer to the "Section 7.14 Prohibited Concomitant Treatments" in the protocol and the corresponding drug washout period regulations.
* Willing and able to complete the planned study assessments, including endoscopic examinations and daily diary records.

Exclusion Criteria:

* Presence of other coexisting autoimmune diseases that may significantly interfere with the attribution of study disease activity or pose additional safety risks. However, if the subject's condition has been clinically stable for ≥ 3 months and is not expected to interfere with study assessments, enrollment may be permitted after confirmation by the investigator and the sponsor's medical monitor (or their designee).

Subjects with the following cardiac diseases will be excluded:

History of heart failure classified as New York Heart Association (NYHA) Class III or IV.

History of myocardial infarction, cardiovascular angioplasty or stenting, unstable angina, or other severe cardiac diseases within 12 months before enrollment.

History of severe central nervous system (CNS) diseases that may affect the subject's ability to comply with the study protocol or interfere with the accuracy of study assessments, such as traumatic brain injury, disturbance of consciousness, epilepsy, cerebral ischemia, or cerebral hemorrhage.

History of malignant tumors other than cured non-melanoma skin cancer or carcinoma in situ (e.g., carcinoma in situ of the cervix, bladder, or breast), unless the subject has been disease-free for at least 3 years.

Primary immunodeficiency. Presence of uncontrolled infection; simple urinary tract infections and upper respiratory tract infections are permitted as judged by the investigator and the sponsor's medical monitor (or their designee).

Known history of infection with human immunodeficiency virus (HIV), hepatitis C virus, or syphilis.

Active or latent hepatitis B virus infection. Positive results for Epstein-Barr virus (EBV) or cytomegalovirus (CMV) DNA or IgM antibodies at screening.

History of recurrent tuberculosis or known presence of recurrent tuberculosis. Subjects with a history of previous chimeric antigen receptor T-cell (CAR-T) therapy or any other genetically modified immune cell therapy will be excluded.

Administration of live-attenuated vaccines within 4 weeks before enrollment. History of allergy to any component of the cell therapy product. History of hypersensitivity to tacrolimus, or previous occurrence of ≥ Grade 3 tacrolimus-related toxicity (including but not limited to neurological, gastrointestinal, hepatic, renal, or hematological toxicity), especially subjects requiring hospitalization, will be excluded. Other cases may be considered eligible after confirmation by the investigator and the sponsor's medical monitor (or their designee).

Participation in another clinical trial within 30 days before screening. Pregnant or lactating subjects, as well as subjects of childbearing potential who cannot use effective contraceptive measures.

Concomitant diseases requiring systemic treatment with therapeutic doses of glucocorticoids (except glucocorticoid treatment for adrenal insufficiency).

Positive results for Clostridioides difficile (C. difficile) toxin or other intestinal pathogens detected within 30 days before colonoscopy screening or at screening. For subjects diagnosed with cytomegalovirus-associated colitis, adequate treatment must be completed and symptoms must be fully resolved for at least 3 months before the screening endoscopy.

Patients with a history of lymphoma, leukemia, or any malignant tumor within the past 10 years are not allowed to enroll.

The following conditions do not exclude enrollment:

Basal cell carcinoma or squamous cell carcinoma of the skin that has been adequately treated with no evidence of metastasis within 1 year; Carcinoma in situ of the cervix that has been adequately treated with no evidence of recurrence within 3 years before baseline.

Patients with significant, uncontrolled neuropsychiatric diseases, patients judged by the investigator to be at risk of suicide, or patients with a history of alcohol dependence and/or substance abuse currently or within the past year are not allowed to enroll.

Presence of unstable or uncontrolled diseases, including but not limited to cerebrocardiovascular, respiratory, gastrointestinal (excluding ulcerative colitis), hepatic, renal, endocrine, hematological, or neurological diseases, which may affect patient safety during the study or interfere with efficacy assessment.

Patients with a known allergy to any component of the investigational drug are not allowed to enroll.

Any other conditions deemed unsuitable for participation in the study by the investigator.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-12-20 (Estimated); Primary Completion 2027-12-30 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events (TEAEs), Serious Adverse Events (SAEs), and Adverse Events of Special Interest (AESIs) | From the day of cell infusion to 24 months after infusion
Serious Adverse Events (SAEs) | Time Frame: From the day of cell infusion to 24 months after infusion
Adverse Events of Special Interest (AESIs) | Time Frame: From the day of cell infusion to 24 months after infusion

SECONDARY OUTCOMES:
Proportion of Patients Achieving Clinical Remission | On the day of cell infusion, and at 28 days, 12 weeks, 24 weeks, 26 weeks, 52 weeks, 76 weeks, and 104 weeks after infusion
Proportion of Patients Achieving Histologic Remission | On the day of cell infusion, and at 28 days, 12 weeks, 24 weeks, 26 weeks, 52 weeks, 76 weeks, and 104 weeks after infusion
Proportion of Patients Achieving Clinical Response | On the day of cell infusion, and at 28 days, 12 weeks, 24 weeks, 26 weeks, 52 weeks, 76 weeks, and 104 weeks after infusion
Proportion of Patients Who Were on Oral Glucocorticoids at Baseline | On the day of cell infusion, and at 28 days, 12 weeks, 24 weeks, 26 weeks, 52 weeks, 76 weeks, and 104 weeks after infusion
Changes in C-Reactive Protein (CRP) | On the day of cell infusion, and at 28 days, 12 weeks, 24 weeks, 26 weeks, 52 weeks, 76 weeks, and 104 weeks after infusion
Achieved Clinical Remission After Treatment Discontinuation of Glucocorticoids | Time Frame: On the day of cell infusion, and at 28 days, 12 weeks, 24 weeks, 26 weeks, 52 weeks, 76
Fecal Calprotectin Levels from Baseline | Time Frame: On the day of cell infusion, and at 28 days, 12 weeks, 24 weeks, 26 weeks, 52 weeks, 76 weeks, and 104 weeks after infusion

CONTACTS AND LOCATIONS:
Overall Officials: Xiaohua Hou, Prof., Principal Investigator — Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Locations (1):
- Union Hospital, Tongji Medical College, Huazhong Univerdity of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No